CLINICAL TRIAL: NCT06212167
Title: The Effect of Nursing Interventions on Stroke Patient Care: Caregivers' Quality of Life, Care Burden, Hopelessness, Anxiety and Depression Levels
Brief Title: Nursing Interventions on Stroke Patient Care: Quality of Life, Hopelessness, Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tuba Yilmaz Bulut, Lecturer Dr., Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-16214662-050.01.04-244840-41
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Depression; Anxiety; Care Burden; Hopefulness
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders; Caregiver Burden | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Interventions for Stroke Patient Care (Experimental): Within the scope of nursing interventions for caregivers;
  * Oral or enteral nutrition application steps and the use of necessary materials will be explained,
  * Oral or enteral drug administration, in-bed exercises, suctioning, simple ROM exercises, in-bed bathing, pressure sore care, position change, oral care, and whole body care will be taught,
  * Videos regarding the use of all medical devices and materials to be taken home with the patient will be shown and demonstration methods will be used,
  * Information about the storage conditions of drugs, side effects and nutrition will be explained, supported by powerpoint presentations,
  * Motivational interviews will be held regarding communication with the stroke patient and the emotional state of the caregivers.
  Interventions: Behavioral: Nursing Interventions for Stroke Patient Care

INTERVENTIONS:
Behavioral: Nursing Interventions for Stroke Patient Care — In the first phase of the research, the relatives of the patients who are in the hospital every day for a week during the routine and discharge process will be included in a training program. These trainings will be explained didactically to the caregiver at the bedside by the research supervisor and the intensive care nurse, the practices will be demonstrated with demonstrations, and the caregiver will be asked to apply them themselves. Then, the researchers will call the caregivers and make an appointment for an online meeting twice a week (7 weeks - 14 times). During these meetings, the training the caregivers need will be explained again and any questions they have will be answered. The researcher will also conduct motivational interviews with the caregivers.

SUMMARY:
In our research, it was aimed to determine the effect of nursing interventions applied face to face at the time of discharge and then via tele-nursing method to the caregivers of patients in intensive care and diagnosed with stroke, on the quality of life, care burden, hopelessness, anxiety and depression levels of the caregivers. This research will be conducted as a randomized, pre-test, post-test single group intervention study, at the Neurology Intensive Care Unit of Sakarya University Training and Research Hospital, between March and June 2023. With a 95% confidence interval, 5% margin of error, 0.54 effect size and 95% representativeness of the population, the group was calculated as 47 people, and the sample was determined as 56 people in total, with 20% reserve. The sample of the study will be selected by simple random sampling method among the caregivers of stroke patients who meet the inclusion criteria and agree to participate in the research. During the discharge process, Information Forms, Zarit Caregiving Burden Scale, Beck Hopelessness Scale, Adult Caregiver Quality of Life Survey, and Hospital Anxiety Depression Scale will be administered face to face to the participants as a pre-test. 12 weeks after the first measurement, Zarit Caregiving Burden Scale, Beck Hopelessness Scale, Adult Caregiver Quality of Life Questionnaire, Hospital Anxiety Depression Scale will be administered as posttest. In addition to routine discharge training, participants will be provided with 'Education and Care Practices for Stroke Patients'. These applications; It will be performed for those who care for stroke patients in the hospital for a week, and then at home, twice a week, for a total of 7 weeks, via telenursing method. Written consent will be obtained from caregivers after explaining the purpose of the research and the purpose for which the results will be used. Participants will be informed that their information will not be shared with others and the confidentiality policy will be adhered to. In order to make comparisons before and after the training, participants will be asked to fill out data collection forms with a nickname they can easily remember and not forget in the pre-test. They will be asked to write the same pseudonyms when filling out the post-test data collection forms. Participants will be asked to fill out data collection forms individually, but it will be stated that they can contact the researchers if they have questions.

ELIGIBILITY:
Inclusion Criteria:

* Having a patient in the Neurology Intensive Care Unit with a diagnosis of stroke,
* The patient is at the stage of being discharged from the intensive care unit,
* Being literate,
* Having a smart phone and being able to use it,
* Having internet access and at least 4GB internet package,
* Volunteering to participate in the research.

Exclusion Criteria:

* Caregivers who are not reachable by phone calls at home,
* Caregivers who do not have continuity in home telenursing training and consultancy practices will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Zarit Caregiving Burden Scale | 1 month
  It was developed by Zarit, Reever and Bach-Peterson in 1980. It is a scale used to evaluate the distress experienced by caregivers of individuals in need of care. The Turkish validity-reliability study of the scale was conducted by İnci and Erdem in 2008. It consists of 22 statements that determine the impact of caregiving on the individual's life. The scale has a Likert-type rating ranging from 1 to 5, such as never, rarely, sometimes, often or almost always. A high scale score indicates that the distress experienced is high. The scoring range is between 0-88, and if the scores obtained are between 0-24 points, "light load"; Between 25 and 33 points is defined as "moderate burden"; Between 34 and 88 points are considered as "severe burden". In the scale form adapted to Turkish, the internal consistency coefficient was found to be 0.95, and the test-retest invariance coefficient was 0.90.
Beck Hopelessness Scale | 1 month
  Beck hopelessness scale was developed by Beck and Weissman (1974). The validity and reliability study of the scale in our country was conducted by Seber, Dilbaz, Kaptanoğlu and Tekin. Durak and Palabıyıkoğlu (1994) conducted a study to examine the validity and factor structure of the scale on a large sample, including physical and psychiatric patients. Beck hopelessness scale consists of 20 true-false situations. 11 of these are correct and 9 are incorrect. Each answer receives 0 or 1 point. The sum of the scores constitutes the despair score. A high score from the scale indicates a high level of hopelessness. Items 1, 6, 13, 15 and 19 describe feelings about the future; Items 2, 3, 9, 11, 12, 16, 17 and 20 describe loss of motivation; Articles 4, 7, 8, 14 and 18 express expectations about the future. Seber et al. (1993), in their hopelessness scale validity and reliability study, determined the Cronbach's alpha coefficient for the entire scale as 0.86.
Adult Caregiver Quality of Life Survey | 1 month
  It is a scale developed by Joseph, Becker, Elwick and Silburn (2012) and its validity and reliability in Turkish was confirmed by Gençer (2020). The scale provides the opportunity to evaluate caregiver quality of life in 8 different areas (caregiving, caregiving preference, patient care stress, financial issues, personal development, appreciation, ability to provide care, and caregiver satisfaction). Each sub-dimension of the scale consists of 5 items. Within forty questions, scoring is applied according to the answers as "Always = 3", "Most of the time = 2", "Sometimes = 1" and "Never = 0", while "6, 7, 8, 9, 10, 11, 12, 13" , 14, 15, 16, 19, 37, 38" questions are coded in reverse (3-2-1-0) and scored. Total score varies between 0-120. 0-40 points indicate "low quality of life", 41-80 points indicate "average quality of life" and 81-120 points indicate "high quality of life". The Adult Caregiver Quality of Life Survey Cronbach's Alpha value was determined as 0.945.
Hospital Anxiety Depression Scale: | 1 month
  Developed by Zigmond and Snaith (1983), hospital anxiety is a four-point Likert type scale consisting of a total of 14 items measuring the level of depression, seven of which (odd numbers) measure anxiety and the other seven (even numbers) measure depression. Aydemir et al. Turkish validity and reliability study was conducted by (1997). Evaluation is made based on the total score. This scale was preferred because it is widely used in both healthy individuals and patients, is easy to apply, and scale scores are not affected by physical symptoms and temporary fluctuations in mood.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University, Kocaeli
  - Sakarya University, Sakarya

IPD SHARING:
Plan to Share IPD: Undecided